CLINICAL TRIAL: NCT02830217
Title: Using Soluble ST2 to Predict Clinical Outcomes in Patients Receiving Primary Percutaneous Coronary Intervention With ST-elevation Myocardial Infarction
Brief Title: Evaluation of Soluble ST2 in Patients Receiving Primary PCI With ST-elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Xuan Zheng, vice director of laboratory of molecular cardiology, Wuhan Asia Heart Hospital
Other Study IDs: 2016LMC-1
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction; Shock
Keywords: STEMI; primary PCI; sST2; prognosis
MeSH Terms: conditions — Myocardial Infarction; Shock; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients having primary PCI: Patients with STEMI receiving primary PCI in Wuhan Aisa Heart Hospital are included in this study. All patients are the first time to have STEMI, and primary PCIs are performed according to 2013 ACCF/AHA guideline for the management of STEMI. Patients with previous stroke, pneumonia, cirrhosis, autoimmune diseases are excluded from this study.

SUMMARY:
ST-elevation myocardial infarction (STEMI) is an urgent symptom associated with sudden myocardial ischemia and ST segment elevated in ECG. Primary percutaneous coronary intervention (PCI) re-open infarct artery efficiently for STEMI patients. However, patients are readmitted shortly after the primary PCI for several unfavorable clinical outcomes including thrombosis in stent, recurrence of myocardial infarction, stroke, and heart failure. This study is intended to test the predictive ability of a new biomarker soluble ST2 (sST2) in peripheral blood. Previous studies have shown that elevated sST2 is highly associated with unfavorable clinical outcomes of patients with ischemia heart diseases and heart failure. This study will further investigate the ability of sST2 to predict unfavorable outcomes for STEMI patients after primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first onset STEMI receive primary PCI according to 2013 ACCF/AHA guideline for management of STEMI

Exclusion Criteria:

* Patients with previous stroke, pneumonia, cirrhosis, autoimmune diseases or severe infection are excluded from this study.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese han population in middle China
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
stent restenosis | one year after primary PCI
  Evidence of stent restenosis of the patients receiving primary PCI, confirmed by coronary angiography when patients are readmitted due to the related symptoms.
recurrence of myocardial infarction | one year after primary PCI
  Evidence of myocardial infarction of the patients receiving primary PCI, confirmed by coronary angiography or ECG when patients are readmitted due to the related symptoms.
heart failure | one year after primary PCI
  Evidence of heart failure of the patients receiving primary PCI, confirmed by clinical diagnosis when patients are readmitted due to the related symptoms.
cardiac death | one year after primary PCI
  Evidence of death due to the cardiac dysfunction of the patients receiving primary PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zheng, MD,PhD, Principal Investigator — Wuhan Asia Heart Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No